CLINICAL TRIAL: NCT05269121
Title: An Open-Label Multicenter Study to Evaluate the Safety and Efficacy of PhageBank™ Phage Therapy in Conjunction With Debridement, Antibiotics, and Implant Retention (DAIR) for Patients With First Time Culture Proven Chronic Prosthetic Joint Infection
Brief Title: Bacteriophage Therapy in First Time Chronic Prosthetic Joint Infections
Acronym: ACTIVE1
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Adaptive Phage Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APT.PJI.002
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Prosthetic Joint Infection; Bacterial Infections
Keywords: Prosthetic; Joint; Knee; Hip; Phage; Bacteriophage; Prosthetic Joint; DAIR
MeSH Terms: conditions — Bacterial Infections | interventions — Phage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DAIR + Phage Treatment + Antibiotics (Experimental): Phage therapy will be administered in conjunction with antibiotics.
  Interventions: Biological: Phage Therapy

INTERVENTIONS:
Biological: Phage Therapy — Patient will undergo a DAIR procedure. After the DAIR, phage therapy will be administered in conjunction with antibiotic treatment.

SUMMARY:
This study will test the feasibility of a regimen of intraoperative (IO) and intravenous (IV) PhageBank™ bacteriophage therapy in conjunction with a DAIR procedure to cure chronic prosthetic joint infection (PJI) without replacement of the prosthesis.

DETAILED DESCRIPTION:
This is a study designed to evaluate bacteriophage therapy in patients with chronic prosthetic joint infections of the hip or knee caused by 1 or 2 of the following organisms: Staphylococcus aureus, Staphylococcus epidermidis, Staphylococcus lugdunensis, Streptococcus spp., Enterococcus faecium, Enterococcus faecalis, Escherichia coli, Pseudomonas aeruginosa, and/or Klebsiella pneumoniae.

This study will compare the safety and efficacy of phage therapy in conjunction with standard of care antibiotics and a DAIR procedure.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥18 years of age.
* Stopped or not received SAT for 2 weeks
* Female patients of childbearing potential who agree to use contraception.
* First time chronic prosthetic joint infection
* Confirmed phage match
* No anticipated need for long-term antibiotics

Exclusion Criteria:

* Soft tissue defect requiring reconstruction.
* Hardware misalignment
* Additional orthopedic hardware in connection with the infected prosthesis.
* Active infection
* Unable to tolerate SAT
* Septic shock or hemodynamic instability.
* Chronic kidney disease
* Liver disease
* Decompensated heart failure.
* Positive drug screen
* Receiving chemotherapy
* Immunocompromised
* Antiviral treatment within 2 weeks prior to DAIR
* Currently participating in another clinical trial
* Known phage allergy
* Pregnant/ breastfeeding
* Lack of capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of phage therapy in adult patients undergoing DAIR for first time chronic prosthetic knee or hip infection | Day 1 through Week 24
  Incidence of reactions to study treatment and discontinuation due to adverse events
Treatment success | 13 months after DAIR
  No recurrence or evidence of infection with the original pathogen at the same joint

SECONDARY OUTCOMES:
No recurrence or evidence of infection for any reason | 3, 6, 13, or 24 months after DAIR
  Infection due to the original or different pathogen at the index site

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hopkins, MD, Study Chair — Adaptive Phage Therapeutics, Chief Medical Officer